CLINICAL TRIAL: NCT04837365
Title: Impact of Neuropsychological Disorders on Visual Exploration, Walking Initiation and Walking in Multiple Sclerosis
Brief Title: Impact of Neuropsychological Disorders in Multiple Sclerosis
Acronym: SEVISEP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lille Catholic University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: RC-P00108
Record Dates: First submitted 2021-04-07; First posted 2021-04-08 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-09

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- patients with neuropsychological disorders (Other)
  Interventions: Other: Three dimensional gait analysis with eyetracking
- patients without neuropsychological disorders (Other)
  Interventions: Other: Three dimensional gait analysis with eyetracking

INTERVENTIONS:
Other: Three dimensional gait analysis with eyetracking — An emotional impregnation and eye pursuit assessment are specific to the study. Emotional impregnation involves making the patient look at images from the International Affective Picture System (IAPS) on a screen before initiating walking. The equipment will be identical to that of the patient during walking tasks. Eye movement analysis is performed using a pair of eyetracking glasses.

SUMMARY:
The study involves MS patients with and without neuropsychological disorders.

The patient will benefit from:

* A routine neuropsychological assessment, including a cognitive and emotional assessment
* A clinical examination
* A three-dimensional analysis of movement

ELIGIBILITY:
Inclusion Criteria:

* Understanding and able to speak French
* Carriers of MS with relapsing remitting form (RRMS-RR) with an EDSS <4
* No significant motor, cerebellar or somesthesia disorders of the upper limbs or visual disturbances (side to a visual EDSS <2)
* Absence of corticosteroid intake in the last four weeks
* Benefiting from health insurance coverage
* Not showing any flare-ups or worsening of the disease in the last 6 weeks
* No botulinum toxin injection for more than 4 months

Exclusion Criteria:

* People with previous neurological pathologies, head trauma with loss of consciousness, psychiatric pathologies, serious general ailments, perceptual or dysarthric disorders preventing verbal communication or reading,
* Treatment with psychotropic drugs (except benzodiazepines and hypnotics).
* Refusal to participate after clear and fair information about the study.
* Adults under tutorship, curatorship or safeguard of justice
* With orthopedic treatment influencing walking
* Pregnant woman

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-05-21 (Actual); Primary Completion 2025-11-21 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Cadence of walking (in cycles.min-1) | 60 days
  The kinematics of the initiation of walking and walking will be appreciated thanks to the variables calculated at the level of the joints of the lower limbs as well as the spatio-temporal parameters without and with management of obstacles (taking a step, balloon)
Step length (in m) | 60 days
  The kinematics of the initiation of walking and walking will be appreciated thanks to the variables calculated at the level of the joints of the lower limbs as well as the spatio-temporal parameters without and with management of obstacles (taking a step, balloon)
Walking speed (in m.s-1) | 60 days
  The kinematics of the initiation of walking and walking will be appreciated thanks to the variables calculated at the level of the joints of the lower limbs as well as the spatio-temporal parameters without and with management of obstacles (taking a step, balloon)
Range of motion in the lower limbs in degrees | 60 days
  The kinematics of the initiation of walking and walking will be appreciated thanks to the variables calculated at the level of the joints of the lower limbs as well as the spatio-temporal parameters without and with management of obstacles (taking a step, balloon)

SECONDARY OUTCOMES:
Ocular fixation time (measured in ms) | 60 days
  Visual exploration will be appreciated by the Ocular fixation time (measured in ms), when initiating walking, walking at spontaneous speed and when passing obstacles with or without a cognitive task. Visual exploration will also be measured after emotional priming when initiating walking and walking. This emotional priming will consist of the transfer of images from the International Affective Picture System (IAPS). This measurement will be carried out using eyetracking glasses worn by patients.
Muscle contractions determined by the electromyogram (EMG) (mV) | 60 days
  The motor patterns (organizations of muscle contractions determined by measuring the EMG of muscles representative of walking) (mV) of the femoral, semi-tendinous, anterior tibial and soleus rectus muscles will be measured using surface EMG , for the two locomotor tasks (walking and initiation to walking), during walking at spontaneous speed (without double task, without crossing an obstacle).
Displacements (in mm) during walking | 60 days
  The displacements (in mm) of the center of the body mass and of the center of pressure on the anteroposterior and mediolateral axes will be derived from the force platforms during the initiation of walking in different conditions (without and with emotional priming).
Acceleration (in mm.s-2) during walking | 60 days
  The acceleration (in mm.s-2) of the center of the body mass and of the center of pressure on the anteroposterior and mediolateral axes will be derived from the force platforms during the initiation of walking in different conditions (without and with emotional priming).
Joint angles | 60 days
  The articular moments and torques (Nm) at the joints of the lower limbs during the initiation to walking will be calculated from kinematic data from the motion analysis laboratory and dynamics of force platforms (without and with priming emotional).

CONTACTS AND LOCATIONS:
Overall Officials: Caroline Massot, MD, Study Director — GHICL
Locations (3):
- France (3):
  - St Vincent hospital - neurological service, Lille
  - St Philibert hospital - Neurologial service, Lomme
  - St Philibert hospital - Physical Medicine and Rehabilitation, Lomme

IPD SHARING:
Plan to Share IPD: No